CLINICAL TRIAL: NCT07225569
Title: A Randomized, Double-blind, Placebo-controlled, Phase 2, Dose-finding Study to Investigate the Efficacy and Safety of SAR445399 in Participants With Moderate to Severe Hidradenitis Suppurativa
Brief Title: A Study to Investigate Efficacy and Safety With SAR445399 in Adult Participants With Moderate to Severe Hidradenitis Suppurativa
Acronym: CLAROS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DRI20674; 2025-522695-83-00 (Registry Identifier: CTIS); U1111-1322-6148 (Other: WHO-ICTRP)
Record Dates: First submitted 2025-11-04; First posted 2025-11-06 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Hidradenitis Suppurativa
MeSH Terms: conditions — Hidradenitis Suppurativa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: [Specify Complex Masking]
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- SAR445399 dose regimen A (Experimental): Participants will receive SAR445399 dose regimen A.
  Interventions: Drug: SAR445399
- SAR445399 dose regimen B (Experimental): Participants will receive SAR445399 dose regimen B.
  Interventions: Drug: SAR445399
- Placebo (Placebo Comparator): Participants will receive SAR445399-matching placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SAR445399 — Pharmaceutical form: Solution for injection/infusion -Route of administration: Injection/infusion
  Arms: SAR445399 dose regimen A; SAR445399 dose regimen B
Drug: Placebo — Pharmaceutical form: Solution for injection -Route of administration: Injection/infusion
  Arms: Placebo

SUMMARY:
This is a multinational, randomized, double-blind, placebo-controlled, Phase 2, dose finding study to evaluate the efficacy and safety of different doses of SAR445399 in adult participants with moderate to severe hidradenitis suppurativa.

The purpose of this study is to assess the efficacy and safety of two doses of SAR445399 compared with placebo in adult participants with moderate to severe hidradenitis suppurativa.

The study duration (per participant) will be up to 30 weeks with a total of 12 visits. The treatment duration will be 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all of the following criteria apply:

* Participants with a history of signs and symptoms consistent with hidradenitis suppurativa (HS) for at least 6 months prior to Baseline
* Participants must have HS lesions present in at least 2 distinct anatomic areas (eg, left, and right axilla; or left axilla and left inguino-crural fold), with at least 1 body site being Hurley Stage II or III.
* Participant must have a total abscess and inflammatory nodule (AN) count of ≥5 at the Baseline Visit.
* Participant must have had an inadequate response to a trial of an oral antibiotic for treatment of HS, exhibited recurrence after discontinuation of antibiotics or demonstrated intolerance to antibiotics or has a contraindication to oral antibiotics for treatment of their HS as assessed by the Investigator through participant interview and review of medical history.
* Participants in the biologic-naïve stratum must be naïve to any prior use of biologic therapy with a potential impact on HS; Participants in the biologic-experienced stratum must have documented history of use of at least one dose of biologic therapy for HS.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* Any other active skin disease or condition (eg, bacterial, fungal, or viral infection) that may interfere with assessment of HS.
* History of recurrent or recent serious infection
* Known history of or suspected current immunosuppression
* History of solid organ transplant or stem cell transplant.
* History of splenectomy
* History of malignancy or lymphoproliferative disease other than adequately treated or nonmetastatic squamous cell carcinoma of the skin that was excised and completely cured or nonmetastatic basal cell carcinoma of the skin that was excised and completely cured.
* Any other medical condition or severe, concomitant illness, including psychiatric illness and substance abuse, that may present an unreasonable risk to the study participants, make participants unreliable or may interfere with study assessments

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2025-12-29 (Actual); Primary Completion 2027-09-22 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants achieving Hidradenitis Suppurativa Clinical Response 75 (HiSCR75) | Up to Week 16
  Hidradenitis Suppurativa Clinical Response 75 (HiSCR75) is defined as ≥75% reduction from baseline in the total abscess and inflammatory nodule [AN] count, with no increase from Baseline in abscess or draining tunnel count.

SECONDARY OUTCOMES:
Percentage of participants achieving Hidradenitis Suppurativa Clinical Response 50 (HiSCR50) | Up to Week 16
  Hidradenitis Suppurativa Clinical Response 50 (HiSCR50) is defined as ≥50% reduction from baseline in the total AN count, with no increase from baseline in abscess or draining tunnel count)
Absolute change from baseline to Week 16 in International Hidradenitis Suppurativa Severity Score System (IHS4) | From baseline to Week 16
  The determination of IHS4 requires counting the inflammatory nodules, abscesses and draining tunnels and multiplying each by a specific coefficient. A high score signifies severe disease.
Percentage of participants achieving Hidradenitis Suppurativa Clinical Response 90 (HiSCR90) | Up to Week 16
  Hidradenitis Suppurativa Clinical Response 90 is defined as ≥90% reduction from baseline in the total abscess and inflammatory nodule [AN] count, with no increase from Baseline in abscess or draining tunnel count.
Percent change from baseline to Week 16 in draining tunnel count | From Baseline to week 16
Absolute change from baseline to Week 16 in draining tunnel count | From Baseline to week 16
Percentage of participants with improvement from baseline to Week 16 of >=3 points in weekly average HS-Skin Pain NRS item 1 from HS-SAQ, among participants with baseline HS-Skin Pain NRS ≥3 | From baseline to Week 16
  The Hidradenitis Suppurativa Symptom Assessment Questionnaire (HS-SAQ) is a 7-item scale comprising unidimensional numeric rating scale (NRS) items assessing symptoms of HS. Hidradenitis Suppurativa Skin Pain Numeric Rating Scale (HS-Skin Pain NRS) is based on worst skin pain in a 24-hour recall period (daily assessment is averaged over 7-day period).
Percent change from baseline to Week 16 in Hidradenitis Suppurativa Skin Pain Numeric Rating Scale (HS-Skin Pain NRS) | From Baseline to Week 16
Absolute change from baseline to Week 16 in the Dermatology Life Quality Index (DLQI) score | From Baseline to Week 16
  The Dermatology Life Quality Index (DLQI) is a 10-item dermatology specific health related quality of life (HRQoL) instrument. Total score ranges from 0 to 30, with higher scores indicating greater detrimental impact on QoL.
Absolute change from baseline to Week 16 in the total Hidradenitis Suppurativa Quality of Life (HiSQoL) score | From Baseline to Week 16
  The Hidradenitis Suppurativa Quality of Life (HiSQoL) is a 17-item content-validated questionnaire with a 7-day recall period. It is scored by summing items to create a total score (0 to 68) with higher score indicating more severe impact on QoL.
Change from baseline to Week 16 in Weekly average HS-SAQ score items | From Baseline to Week 16
  The Hidradenitis Suppurativa Symptom Assessment Questionnaire (HS-SAQ) is a 7-item scale comprising unidimensional numeric rating scale (NRS) items assessing symptoms of HS. Each item is scored on a 0 to 10 scale with 0 indicating "no symptom" and 10 indicating "worst symptom possible".
Change from baseline to Week 16 in the Hidradenitis Suppurativa Impact Assessment Questionnaire (HS-IAQ) score | From Baseline to Week 16
  The Hidradenitis Suppurativa Impact Assessment Questionnaire (HS-IAQ) is an 11-item questionnaire assessing the impact of HS on QoL
Improvement in Peak Pruritus Numerical Rating Scale (PP-NRS) at Week 16 | From Baseline to Week 16
  The Peak Pruritus Numerical Rating Scale (PP-NRS) is defined as achieving at least 4-unit reduction from Baseline in weekly average of daily PP-NRS among participants with baseline PP-NRS ≥4)
Number of participants with Treatment Emergent Adverse Events (TEAEs) Adverse Events of Special Interest (AESIs), and Serious Adverse Events (SAEs) including administration site reactions | Up to End of Study (approximately 30 weeks)
Number of participants with potentially clinically significant abnormalities in laboratory tests, vital signs, and electrocardiograms (ECGs) | Up to End of Study (approximately 30 weeks)
Serum concentrations of SAR445399 throughout the study | Up to End of Study (approximately 30 weeks)
Incidence of anti-drug antibodies (ADA) of SAR445399 at prespecified timepoints | Up to End of Study (approximately 30 weeks)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (3):
  - Carbon Health - North Hollywood - NoHo West- Site Number : 8400017, North Hollywood, California
  - Florida International Research Center- Site Number : 8400002, Miami, Florida
  - Equity Medical- Site Number : 8400010, New York, New York
- Investigational Site Number : 1560001, Beijing, China
- Investigational Site Number : 3480001, Debrecen, Hungary

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: DRI20674 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=26984&tenant=MT_SNY_9011